CLINICAL TRIAL: NCT06460545
Title: Phase IV Study of Evaluating Immunogenicity and Safety of Concomitant Administration of Sabin-strain-based Inactivated Poliovirus Vaccine (Vero Cells) and Freeze-dried Live-attenuated Hepatitis A Vaccine or Inactivated Hepatitis A Vaccine
Brief Title: Phase IV Study of Concomitant Administration of the sIPV and HepA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sIPV-402
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Polio; Hepatitis A
MeSH Terms: conditions — Poliomyelitis; Hepatitis A | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- sIPV + HepA-L (coconmitant vaccination cohort) (Experimental): Concomitant administration of sIPV and HepA-L at 18 months of age
  Interventions: Biological: sIPV (booster dose at 18 months of age); Biological: HepA-L
- sIPV + HepA-I (coconmitant vaccination cohort) (Experimental): Concomitant administration of sIPV and HepA-I at 18 months of age, and another dose administration of HepA-I at 24 months of age
  Interventions: Biological: sIPV (booster dose at 18 months of age); Biological: HepA-I
- sIPV (individual vaccination cohort) (Experimental): One booster dose of sIPV at 18 months of age
  Interventions: Biological: sIPV (booster dose at 18 months of age)
- HepA-L (individual vaccination cohort) (Experimental): One dose of Hep-L at 18 months of age
  Interventions: Biological: HepA-L
- HepA-I (individual vaccination cohort) (Experimental): Two doses of Hep-I at 18 and 24 months of age, respectively
  Interventions: Biological: HepA-I

INTERVENTIONS:
Biological: sIPV (booster dose at 18 months of age) — Sabin-strain-based inactivated vaccine (Vero cells), 0.5mL for each dose at 18 months of age for the booster one
  Arms: sIPV (individual vaccination cohort); sIPV + HepA-I (coconmitant vaccination cohort); sIPV + HepA-L (coconmitant vaccination cohort)
Biological: HepA-L — Freeze-dried/lyophilized live-attenuated hepatitis A virus vaccine, 1.0mL for each dose at 18 months of age
  Arms: HepA-L (individual vaccination cohort); sIPV + HepA-L (coconmitant vaccination cohort)
Biological: HepA-I — Inactivated hepatitis A virus vaccine, 0.5mL for each dose, two doses at 18 and 24 months of age, respectively
  Arms: HepA-I (individual vaccination cohort); sIPV + HepA-I (coconmitant vaccination cohort)

SUMMARY:
This study is a randomized, open-labeled phase IV clinical trial to evaluate the immunogenicity and safety of concomitant administration of sIPV and HepA-L or HepA-I in children aged 18 months. The primary immunogenicity endpoints in all groups are the seroconversion rates of type I, II, and III anti-poliovirus neutralizing antibodies and the seroconversion rate of anti-hepatitis A virus antibodies 30 days after the final administration. The secondary immunogenicity endpoints are (1) the GMT/GMC of type I, II, and III anti-poliovirus neutralizing antibodies as well as the anti-hepatitis A virus antibodies 30 days after the final administration; (2) the seropositive rates of the anti-hepatitis A virus antibodies 30 days after the final administration; (3) the GMFI of type I, II, and III anti-poliovirus neutralizing antibodies as well as the anti-hepatitis A virus antibodies 30 days after the final administration. The secondary safety endpoints are the incidence of adverse events (AEs) within 30 minutes after each injection, the incidence of solicited local and systematic AEs in the period of solicitation after each injection, the incidence of unsolicited AEs in 30 days after each injection, the incidence of AEs in 30 days after each injection, and the incidence of serious adverse events in 6 months after administrations.

DETAILED DESCRIPTION:
This is a randomized, open-labeled, parallel phase IV clinical trial to evaluate the immunogenicity and safety of concomitant administration of sIPV and HepA-L or HepA-I. 2000 children subjects aged 4 months will be enrolled to take administration of 1 dose of sIPV. All participants at 18 months of age will be randomly assigned to 5 cohorts in a ratio of 4:4:4:3:3, that is, (1) 400 subjects will be concomitantly injected with sIPV and HepA-L, (2) 400 subjects will be concomitantly injected with sIPV and HepA-I, and another dose of HepA-I at 24 months of age (3) 400 subjects will be only injected one dose of sIPV, (4) 300 subjects will be only injected with one dose of HepA-L, (5) 300 subjects will be only injected with two doses of HepA-I at 18 and 24 months of age, respectively.

For safety assessment, adverse events after the third dose of sIPV at 4 months of age would be collected through phone-call follow-ups on Day 8 and Day 30 after the injection by investigators and active reports from participants' guardians. At 18 months of age, safety data would be recorded through the diary and contact cards by participants' guardians to collect solicited or unsolicited AEs in periods of solicitation and nonsolicitation, respectively. From 31 days after the final dose to 6 months later, serious adverse events will be evaluated by the investigator via phone call or active reports by participants' guardians.

For immunogenicity assessment, blood samples before each dose on Day 0 and Day 30 after each injection would be collected to evaluate the type I, II, and III anti-poliovirus neutralizing antibody levels or/and anti-hepatitis A virus antibody for different groups.

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: Children aged 4 months at the time of enrollment
* Vaccination Requirement: volunteers have already taken administration 2 doses of sabin-strain-based inactivated poliovirus vaccine (produced by IMBCAMS), and have not yet been injected with the third dose containing poliovirus antigen.
* Provision of Legal Identification: Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Informed Consent: Legal guardians or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, and sign the informed consent form.
* Adherence: Legal guardians or appointed representatives of volunteers must be able to comply with the requirements in the study as well as complete relevant visits on time.
* Birth condition: Full-term birth (37~42 gestational weeks) and normal birth weight (no less than 2500g).
* Temperature Requirement: Axillary body temperature prior to vaccination is less than 37.3°C.

Exclusion Criteria:

* Health Requirement: Volunteers cannot meet health requirements through physical examinations.
* History of Related Illness: Volunteers have a history of developing Hepatitis A, poliomyelitis, or immunodeficiency.
* Birth Condition: Volunteers have a history of abnormal labor stage, asphyxia, nervous system damage, or clinically confirmed pathologic jaundice。
* Allergic History: Volunteers have a history of allergies to any component of the investigational vaccine (e.g., aluminum hydroxide), any history of vaccine allergies, suspected allergies, or any other severe adverse reactions.
* Vaccine History: Volunteers received any inactivated vaccines or subunit vaccines within 7 days (including the 7th day) prior to vaccination with the investigational vaccine, or any other live attenuated vaccines within 14 days (including the 14th day) prior to vaccination.
* Acute Illness: Volunteers have experienced acute illnesses (e.g., fever) within 3 days prior to vaccination with the investigational vaccine.
* Neurological and Mental Health: Volunteers have a history of seizures, convulsions, cerebral palsy, epilepsy, mental illness, or a family history of such conditions.
* Health Conditions: Volunteers have known congenital abnormalities, developmental disorders, genetic defects, or severe malnutrition, among other conditions.
* Coagulation Abnormalities: Volunteers have a history of coagulation disorders (e.g., coagulation factor deficiency, coagulation disorders).
* Infectious Diseases: Volunteers have infectious diseases that may affect the study, such as human immunodeficiency virus (HIV) infection, hepatitis, and tuberculosis.
* Special Condition: Volunteers who could not tolerate venipuncture, or had a history of needle and blood sickness.
* Organ Removal History: Volunteers have a history of organ removal (e.g., thyroid, pancreas, liver, spleen).
* History of Blood Products: Volunteers have a history of loss of blood, blood transfusion, the use of adjuvant therapies, or immunoglobulin within 3 months prior to vaccination.
* Immune Therapy: Volunteers have received immune-enhancing or immune-suppressing therapy within the last 3 months (continuous oral or intravenous administration for more than 14 days) prior to vaccination.
* Participation in Other Clinical Studies: Volunteers are currently or have plans to participate in other clinical studies before enrollment.
* Investigator's Discretion: The final exclusion criterion is the investigator's discretion to determine whether a volunteer is suitable for participation in the study.

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-seroconversion rate of type I anti-poliovirus neutrilizing antibody | Between baseline and day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of type II anti-poliovirus neutrilizing antibody | Between baseline and day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline
Immunogenicity index-seroconversion rate of type III anti-poliovirus neutrilizing antibody | Between baseline and day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline
Immunogenicity index-seropositive rate of type I anti-poliovirus neutrilizing antibody | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as the level (≥1:8).
Immunogenicity index-seropositive rate of type II anti-poliovirus neutrilizing antibody | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as the level (≥1:8).
Immunogenicity index-seropositive rate of type III anti-poliovirus neutrilizing antibody | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method. Seroconversion will be defined as the level (≥1:8).
Immunogenicity index-seroconversion rate of anti-hepatitis A virus antibody | Between baseline and day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<20mIU/ml) to seropositive (≥20mIU/ml), or a ≥4-fold increase from baseline

SECONDARY OUTCOMES:
Immunogenicity index-geometric mean titer (GMT) of type I anti-poliovirus neutrilizing antibody | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type II anti-poliovirus neutrilizing antibody | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean titer (GMT) of type III anti-poliovirus neutrilizing antibody | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean concentration (GMC) of anti-hepatitis A virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Immunogenicity index-seropositive rate of anti-hepatitis A virus antibody | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the level (≥20mIU/ml).
Immunogenicity index-geometric mean fold increase (GMFI) of type I anti-poliovirus neutrilizing antibody | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type II anti-poliovirus neutrilizing antibody | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of type III anti-poliovirus neutrilizing antibody | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization method.
Immunogenicity index-geometric mean fold increase (GMFI) of anti-hepatitis A virus antibody | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method.
Safety index-incidence of adverse events | 0-30 minutes after vaccination
  Incidence of adverse events after vaccination
Safety index-incidence of solicited adverse events | Day 0-7 or Day 0-14 after vaccination
  Incidence of solicited local and systematic adverse events after vaccination
Safety index-incidence of unsolicited adverse events | Day 0-30 after vaccination
  Incidence of unsolicited adverse events after vaccination
Safety index-incidence of adverse events | Day 0-30 after vaccination
  Incidence of adverse events after vaccination
Safety index-incidence of serious adverse events | From the beginning of the vaccination up to 6 months after vaccination completed
  Incidence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jiawei Xu, Principal Investigator — Chongqing Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Jiu Longpo District Center for Disease Control and Disease, Chongqing, Chongqing Municipality
  - Wanzhou District Center for DIsease Control and Prevention, Chongqing, Chongqing Municipality
  - Jiangjin District Center for Disease Control and Prevention, Chongqing, Chonqing

IPD SHARING:
Plan to Share IPD: No